CLINICAL TRIAL: NCT03363711
Title: AYA STEPS RCT: AYA Self-Management Via Texting, Education & Plans for Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 26916
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Adolescent and Young Adult (AYA) Cancer Survivors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AYA STEPS — a mobile health application

SUMMARY:
The proposed project will leverage two programs of research at UPenn and CHOP that are delivering technology-based interventions to adolescent and young adult (AYA) cancer survivors.

In the proposed study, all AYA survivors will receive a care plan via a tool (Smart-ALACC). They will then be randomized to receive (or not) a mobile health application (AYA STEPS) that will provide tailored messages to enhance uptake of their care plan.

ELIGIBILITY:
Inclusion Criteria:

* AYA is 15-29 year old with a history of a malignant cancer diagnosis;
* Completed cancer treatment and are currently in remission or receiving cancer survivorship care;
* Seen for follow-up oncology care at CHOP or Penn;
* For AYA less than 18 years old, must have a caregiver to provide informed consent.

Exclusion Criteria:

* Cognitive impairments that would limit AYA ability to independently care for health as determined by the medical team.
* Absence of the inclusion criteria

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 15-29 year olds with a history of malignant cancer diagnosis.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Completed mobile data and questionnaires | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine Hill-Kayser, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Psihogios AM, King-Dowling S, O'Hagan B, Darabos K, Maurer L, Young J, Fleisher L, Barakat LP, Szalda D, Hill-Kayser CE, Schwartz LA. Contextual Predictors of Engagement in a Tailored mHealth Intervention for Adolescent and Young Adult Cancer Survivors. Ann Behav Med. 2021 Nov 18;55(12):1220-1230. doi: 10.1093/abm/kaab008. PMID 33674863